CLINICAL TRIAL: NCT01679691
Title: The Effect of Epidural Anesthesia on the Intra-operative and Post-operative Amount of Bleeding Following Lower Limb Salvage Surgery
Brief Title: The Epidural Anesthesia on the Intra-operative and Post-operative Amount of Bleeding Post Lower Limb Salvage Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Till IRB renewal
Sponsor: Children's Cancer Hospital Egypt 57357 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CCHE-BoneT001
Record Dates: First submitted 2012-08-12; First posted 2012-09-06 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Bone Tumor
MeSH Terms: conditions — Bone Neoplasms | interventions — Anesthesia, Epidural

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (No Intervention): Control group in whom no epidural anesthesia will be applied
- Epidural Anesthesia (Active Comparator): the group in whom all patients will be subjected to epidural anesthesia intra- and post-operative
  Interventions: Other: epidural anesthesia

INTERVENTIONS:
Other: epidural anesthesia — the group in whom all patients will be subjected to epidural anesthesia intra- and post-operative
  Arms: Epidural Anesthesia

SUMMARY:
Epidural anesthesia is a very useful tool in lower limb salvage surgery, which helps pain control intra and more importantly post-operative pain. It is a well-known effect of epidural injections to cause a sympathetic stimulation and consequently vasodilatation in the lower limb vessels.

Since epidural catheters can cause vasodilatation in lower limb vessels, they can subsequently lead to increased intra and post-operative bleeding from the surgical wound.

The study will involve all patients having a bone tumor in the lower limb and subjected to tumor resection and reconstruction by prosthesis.

The patient will be randomized according to the administration of epidural anesthesia into two arms, an arm in which epidural anesthesia was employed and another arm in which the patient was subjected only to general anesthesia and the amount of intra and postoperative bleeding will be compared in both arms.

DETAILED DESCRIPTION:
Assessment of intra-operative bleeding will be based upon weighing and counting of the blood soaked dressing and the amount of blood transfusion used.

Assessment of post-operative bleeding will be based upon the amount of blood collected from the suction drain and amount of blood transfusion.

All patient subjected to anticoagulant post-operative or another type of surgery other than implantation of prosthesis will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* lower limb bone tumor
* reconstruction by prosthesis

Exclusion Criteria:

* upper limb and pelvic salvage surgery.
* other methods of reconstruction than prosthesis
* use of tourniquet intra-operative.
* post-operative anticoagulation.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2011-09; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Measure the blood loss intra- and post-operative in both the contro and study groups | start of surgery until removal of sucction drain
  The amount of blood loss will be assessed using:
  * Intra-operative: measurement of dressing before and after being soaked.
  * Post-operative: amount of blood drainage and duration of use of the suction drain.

SECONDARY OUTCOMES:
prolongation of hospital stay | the number of days calculated from date of surgery until dischare from hospital expected average from 5 to 7 days
  the number of days calculated from date of surgery until discharge from hospital expected average from 5 to 7 days

CONTACTS AND LOCATIONS:
Overall Officials: ahmed elghoneimy, MD, Principal Investigator — Children's Cancer Hospital Egypt 57357
Locations (1):
- Children's Cancer Hospital Egypt-57357, Cairo, Egypt